CLINICAL TRIAL: NCT03096301
Title: Photomodulation in the Treatment of Pain in Patients With Tmd: Analysis of Cost-effectiveness.
Brief Title: Photobiomodulation in Temporomandibular Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Lara Jansiski Motta, Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CEPhotobio01
Record Dates: First submitted 2017-03-09; First posted 2017-03-30 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Pain; Temporomandibular Disorder
Keywords: temporomandibular disorder; photobiomodulation; pain
MeSH Terms: conditions — Pain; Temporomandibular Joint Disorders

STUDY DESIGN:
Intervention Model Description: It is a prospective trial of clinical and economic analysis. It will include 45 patients to evaluate the effectiveness of the treatments with low-intensity laser and occlusal plate for muscle pain in patients with TMD
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-intensity laser (Experimental): Twelve laser applications will be applied as initial treatment, with 2 sessions per week. A wave length of 780 nm, with an energy density of 25 J/cm2, a power of 50 mW and power density of 1.25 W/cm2, will be used for a duration of 20 seconds per point, resulting in a total energy of 1J per point. The laser will be applied at each point, using a conventional tip in contact with the skin, thus considering an area of 0.04 cm2, in accordance with the protocol suggested by Venezian et al. (2010) and Carvalho et al. (2010). The laser will be applied to 3 points of the masseter muscle (upper, middle, and lower bundles) and 1 point in the anterior temporalis on each side of the face
  Interventions: Device: Low-intensity laser; Device: Placebo
- Occlusal Plate (Active Comparator): The group undergoing treatment with occlusal plates will be instructed to use the device during sleep, 8 hours per night, for a period of 12 months. The plates will be made following the principles established by Okenson (1998).
  Participants will be molded with alginate to obtain models. In the upper model, a 2 mm acetate plate will be made, to be later replaced with acrylic resin (STRINI et al., 2009), and these plates will be adjusted in centric relation, to promote occlusal stability and disocclusion guide.
  Weekly follow-up and adjustments will be performed during the evaluation period, until the completion of treatment
  Interventions: Device: occlusal plates; Device: Placebo
- Placebo (Placebo Comparator): For the placebo group, all the measures described for the group 1 (LIL) will be adopted, however the laser equipment will remain switched off.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Low-intensity laser — Laser applications will be applied as initial treatment, with 2 sessions per week. A wave length of 780 nm, with an energy density of 25 J/cm2, a power of 50 mW and power density of 1.25 W/cm2, will be used for a duration of 20 seconds per point, resulting in a total energy of 1J per point. The laser will be applied at each point, using a conventional tip in contact with the skin, thus considering an area of 0.04 cm2
  Arms: Low-intensity laser
Device: occlusal plates — The group undergoing treatment with occlusal plates will be instructed to use the device during sleep, 8 hours per night, for a period of 12 months. The plates will be made following the principles established by Okenson (1998).
  Participants will be molded with alginate to obtain models. In the upper model, a 2 mm acetate plate will be made, to be later replaced with acrylic resin (STRINI et al., 2009), and these plates will be adjusted in centric relation, to promote occlusal stability and disocclusion guide.
  Weekly follow-up and adjustments will be performed during the evaluation period, until the completion of treatment
  Arms: Occlusal Plate
Device: Placebo — For the placebo group, all the measures described for the group 1 (LIL) will be adopted, however the laser equipment will remain switched off.

SUMMARY:
The general purpose of this project is to evaluate the cost-effectiveness of LIL treatment and occlusal plates in the treatment of pain in patients between 15 and 25 years of age with TMD.

DETAILED DESCRIPTION:
Temporomandibular disorder (TMD) affects a significant portion of the population. Epidemiological data show that the signs and symptoms of TMD start to become apparent from six years of age, and in adolescence these signs and symptoms are similar to those of adults. The painful conditions of TMD can affect the quality of life of young patients, compromising the daily activities of these individuals. The present project aims (1) to estimate the direct costs of treatment of muscle pain in patients with TMD with low-intensity laser and with occlusal plate and a placebo group; (2) to evaluate the effectiveness of the treatments with low-intensity laser and occlusal plate for muscle pain in patients with TMD; (3) to analyze the cost-effectiveness of the two proposed treatments for pain; and (4) to describe and compare the results of analyses of treatments for pain in patients with TMD. The study will be conducted at the Odontological Clinic of Universidade Nove de Julho. It is a prospective trial of clinical and economic analysis. It will include 30 patients aged between 15 and 25 years with TMD, randomly assigned to a treatment group: G1 (low-power laser), G2 (occlusal plate) and G3 (placebo). The analysis will be based on the direct costs of each treatment during the 12-month period, estimating the cost of each treatment. The outcome for the analysis of the effectiveness will be the pain, measured periodically by means of the clinical examination of the Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD). The cost-effectiveness ratio will be calculated using, as endpoints, pain and the calculation of the ratio between the difference in costs between the groups studied. The evaluation of the impact of the treatment on quality of life will be determined by applying the adapted EuroQol-5D.

ELIGIBILITY:
Inclusion Criteria:

* people between 15 and 25 years
* diagnosis of TMD in group I

Exclusion Criteria:

* Individuals with dental-facial anomalies
* orthodontic or orthopedic treatment
* Individuals who were taking muscle relaxants or anti-inflammatory medications

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-01-21 (Actual); Study Completion 2018-10-10 (Estimated)

PRIMARY OUTCOMES:
Pain | 12 months after treatment
  Muscle pain will be analyzed by clinical criteria of the Research Diagnostic Criteria for Temporomandibular Disorders

SECONDARY OUTCOMES:
Cost-effectviness | 12 months after treatment
  This phase of the study will consist in the quantification of resources, i.e. determining the frequency of use of resources and materials during the treatment. The units used to quantify the direct costs consumed are physical units such as consultation time, number of sessions, equipment used, and materials consumed. These data will be collected using a specific form.

CONTACTS AND LOCATIONS:
Locations (1):
- Lara Motta, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sobral APT, Godoy CLH, Fernandes KPS, Bussadori SK, Ferrari RAM, Horliana ACRT, Monken SF, Motta LJ. Photomodulation in the treatment of chronic pain in patients with temporomandibular disorder: protocol for cost-effectiveness analysis. BMJ Open. 2018 May 5;8(5):e018326. doi: 10.1136/bmjopen-2017-018326. PMID 29730613